CLINICAL TRIAL: NCT06718543
Title: A Multicenter, Randomized, Parallel, Non-Controlled, Prospective Phase II Study of Neoadjuvant Short-Course Radiotherapy Sequential With AK112 With or Without Chemotherapy for Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Short-Course Radiotherapy With or Without Chemotherapy and AK112 in Locally Advanced Rectal Cancer
Acronym: TRIUNITE-03
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: fan li (Other)
Responsible Party: Sponsor-Investigator, fan li, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIUNITE-03
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; neoadjuvant; Ivonescimab; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCRT followed by CapeOX regimen combined with AK112 (Experimental): Patients will receive short-course radiotherapy (SCRT) followed by chemotherapy (CapeOX regimen) combined with AK112:
  In the 1st week, neoadjuvant short-course radiotherapy will be administered (25 Gy in 5 fractions over 5 days). After a 7-day interval, patients will receive 2 cycles of CapeOX chemotherapy combined with AK112 (every 3 weeks; Day 1: Oxaliplatin, 130 mg/m², IV infusion; Day 1: AK112, 20 mg/kg, IV infusion; Day 1 to Day 14: Capecitabine, 850-1000 mg/m², BID, orally).
  Interventions: Drug: AK112 with SCRT and CapeOX
- SCRT followed by AK112 (Experimental): Patients will receive short-course radiotherapy (SCRT) followed by AK112:
  In the 1st week, neoadjuvant short-course radiotherapy will be administered (25 Gy in 5 fractions over 5 days). After a 7-day interval, patients will receive 2 cycles of AK112 treatment (Day 1: AK112, 20 mg/kg, IV infusion).
  Interventions: Drug: AK112 with SCRT

INTERVENTIONS:
Drug: AK112 with SCRT and CapeOX — In the 1st week, neoadjuvant short-course radiotherapy will be administered (25 Gy in 5 fractions over 5 days). After a 7day interval, patients will receive 2 cycles of CapeOX chemotherapy combined with AK112 (every 3 weeks; Day 1: Oxaliplatin, 130 mg/m², IV infusion; Day 1: AK112, 20 mg/kg, IV infusion; Day 1 to Day 14: Capecitabine, 850-1000 mg/m², BID, orally).
  Other Names: short-course radiotherapy; CapeOX
  Arms: SCRT followed by CapeOX regimen combined with AK112
Drug: AK112 with SCRT — In the 1st week, neoadjuvant short-course radiotherapy will be administered (25 Gy in 5 fractions over 5 days). After a 7-day interval, patients will receive 2 cycles of AK112 treatment (Day 1: AK112, 20 mg/kg, IV infusion).
  Arms: SCRT followed by AK112

SUMMARY:
This phase II multicenter, randomized study evaluates the safety and efficacy of neoadjuvant short-course radiotherapy (SCRT) sequentially combined with AK112 (Envafolimab) with or without chemotherapy in patients with locally advanced rectal cancer (LARC). The study also aims to identify biomarkers predicting tumor response and develop efficacy prediction models.

DETAILED DESCRIPTION:
The study is designed as a two-arm, randomized, open-label, prospective trial. Patients with locally advanced rectal adenocarcinoma will be randomly assigned to one of two treatment groups:

Arm A: SCRT followed by chemotherapy (CapeOX) combined with AK112. Arm B: SCRT followed by AK112 alone. Primary and secondary outcome measures include complete response rate (CR), safety, pathological and radiological response rates, and biomarkers associated with treatment response. The trial will enroll 100 participants across multiple centers over three years.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age 18-80 years, male or female.
3. Histologically confirmed rectal adenocarcinoma.
4. Clinical baseline stage T3-4NxM0 or TxN1-2M0 by MRI assessment.
5. Able to swallow tablets.
6. ECOG Performance Status of 0-1.
7. No prior treatment for rectal cancer, including surgery, radiotherapy, 8.chemotherapy, immunotherapy, or targeted therapy.

9.Fit for surgery with no contraindications. 10.Normal organ function. 11.Tumor ≤12 cm from the anal verge

Exclusion Criteria:

1. Allergy to monoclonal antibodies, AK112 components, or CapeOX regimen.
2. Previous or current use of immune checkpoint inhibitors or immune-related 3.treatments.

4.Active autoimmune diseases or history of significant autoimmune conditions. 5.Immunodeficiency disorders or history of organ/bone marrow transplantation. 6.Uncontrolled cardiovascular conditions (e.g., heart failure, unstable angina, recent MI).

7.Severe infection within 4 weeks or active pulmonary infections. 8.Active hepatitis B or C infection. 9.Diagnosis of other malignancies within 5 years (except low-risk cancers). 10.Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | From treatment initiation to post-neoadjuvant therapy evaluation (approximately 12 weeks).
  Proportion of patients achieving either a pathological complete response (pCR) or a clinical complete response (cCR).

SECONDARY OUTCOMES:
Adverse Events (AEs) | From baseline to 90 days after the last treatment dose.
  Incidence, type, and severity of adverse events graded according to CTCAE v5.0, including their correlation with the study drug.
Major Pathological Response (MPR) | At the time of surgery (approximately 12 weeks after treatment initiation).
  Proportion of patients with ≤10% residual viable tumor cells in resected specimens.
Objective Response Rate (ORR) | Approximately 12 weeks after treatment initiation.
  Proportion of patients with complete response (CR) or partial response (PR) based on radiological assessments using RECIST 1.1 criteria.
Progression-Free Survival (PFS) | Up to 36 months post-randomization.
  Time from randomization to disease progression or death from any cause.
Overall Survival (OS) | Up to 36 months post-randomization.
  Time from randomization to death from any cause.
Organ Preservation Rate (OPR) | Approximately 12 months post-treatment initiation.
  Proportion of patients avoiding major surgery while retaining organ functionality.
Tumor Response Based on RECIST 1.1 | Approximately 12 weeks after treatment initiation.
  Evaluation of complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) using RECIST 1.1 criteria.
Clinical Complete Response Rate (cCR) | Approximately 12 weeks after treatment initiation.
  Proportion of patients achieving clinical complete response based on clinical examination and imaging assessments.
Pathological Complete Response (pCR) | Approximately 12 weeks after treatment initiation.
  Absence of tumor cells in the primary tumor and regional lymph nodes in surgical specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No